CLINICAL TRIAL: NCT01574066
Title: Chest CT-scan for the Diagnosis of Community-acquired Pneumonia in Patients Visiting the Emergency Department
Brief Title: Chest CT-scan for the Diagnosis of Community-acquired Pneumonia
Acronym: PACSCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM10014; P100121 (Other Grant/Funding Number: AP-HP)
Record Dates: First submitted 2012-02-07; First posted 2012-04-10 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Community-acquired Pneumonia; Dyspnea
Keywords: Community-acquired pneumonia; Diagnosis; Emergency medicine; Chest CT-scan
MeSH Terms: conditions — Community-Acquired Pneumonia; Dyspnea; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chest CT-scan (Experimental): Patients with a suspicion of acquired pneumonia visiting the emergency department will do a chest CT-scan
  Interventions: Procedure: Chest CT-scan

INTERVENTIONS:
Procedure: Chest CT-scan — Patients with a suspicion of acquired pneumonia visiting the emergency department will do a chest CT-scan

SUMMARY:
Primary objective : to estimate impact of CT-scan on diagnostic for emergency department (ED) patients with suspected Community-acquired Pneumonia (CAP).

Secondary objective: to estimate impact of CT-scan on treatment (antimicrobial therapy) and site of care for ED patients with suspected CAP.

DETAILED DESCRIPTION:
Rational: Community-acquired pneumonia (CAP) is a frequent infectious disorder in patients visiting the ED. CAP is responsible for high morbidity and associated-mortality is increasing in Western countries. CAP corresponds to invasion of the lung by pathogens. Diagnosis depends on clinical and X-ray assessment. However, these signs and symptoms are poorly specific and are often lacking. As prognosis depends on precocious and fitted antimicrobial treatment, making CAP diagnosis in a short time span (4-8 hours) is mandatory. Preliminary studies suggest that chest CT-scan could over-performed X-ray for diagnosis of CAP. Consensus conferences suggest the use of CT-scan in patients with uncertain diagnosis and unusual presentation and outcome. Because CT-scan is currently easily available, its use in a first intent is questionable for ED patients with suspected CAP.

Primary objective: to estimate impact of CT-scan on diagnostic for ED patients with suspected CAP.

Secondary objective: to estimate impact of CT-scan on treatment (antimicrobial therapy) and site of care for ED patients with suspected CAP.

Prospective multicenter study to measure chest CT-scan impact. 350 patients visiting the ED of 4 inner tertiary teaching hospitals in Paris, France, with suspected CAP.

Management: Patients will be managed according to current guidelines, including conventional chest X-ray.

Evaluation criteria. Attending ED physicians will implement pre- and post-test proforma for diagnosis (CAP) level of certainty, treatment (antimicrobial agents), site of care, before and after chest CT-scan. Comparison of ED physician's answers before/after CT-scan. Patients will be followed until day 28. An adjudication committee (1 pneumologist, 1 infectiologist, 1 radiologist)will review patients' data for gold standard diagnosis.

Statistical considerations: The investigators hypothesize that chest CT-scan wil modify diagnosis certainty in 20%. This implies that 300 participants should be enrolled to allow assessment of changes in 15 % et 25 %. Undue changes will be calculated a posteriori when diagnosis gold standard will be established by adjudication committee.

Anticipated results: Chest CT-scan should improve diagnosis certainty, treatment and site-of-care in patients visiting the ED with suspected CAP. If this is observed in at least 20%, the investigators will measure impact of chest CT-scan in a prospective randomized interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 years of age
* Patient with a presumptive diagnosis of CAP according to attending ED physician
* Patient experiencing at least one systemic sign (T°>38°C or < 36°C, HR>90/min, RR>20/min)
* Patient experiencing one respiratory sign (cough, lateral chest pain, localized crackles, dyspnea) that recently appeared
* Patient with a prior medical examination, the results have been or will be communicated
* Patient gave written informed consent or in cases of emergency parent/ support person who gave written informed consent if he/she is present on the day of inclusion

Exclusion Criteria:

* Pregnancy
* Patient with shock
* Patient with respiratory distress and immune suppression
* Patient with other criteria for immediate ICU referral to ICU
* Patient with living conditions making it impossible to follow 28 days
* Patient not affiliated with a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Chest CT-scan | in 28 days
  Percentage of diagnoses modified by chest CT-scan.

SECONDARY OUTCOMES:
Treatments changes | in 28 days
  Percentage of treatments changes (antimicrobial therapy) modified by chest CT-scan
Changes of site-of-care | in 28 days
  Percentage of site-of-care (admission/non admission) modified by chest CT-scan
Identification of viral and bacterial agents | at day of inclusion (day 1)
  Identification of viral and bacterial agents from nasal and pharyngeal swabs
Markers of infection in the blood | at day of inclusion (day 1)
  Determination of markers of infection in the blood
Markers of infection and markers of inflammation in urine | at day of inclusion (day 1)
  Determination of markers of infection and of inflammation in urine

CONTACTS AND LOCATIONS:
Overall Officials: Yann-Erick Claessens, MD, PhD, Principal Investigator — Cochin Hospital, Paris, France
Locations (4):
- France (4):
  - La Pitié Salpêtrière Hospital, Paris
  - Cochin Hospital, Paris
  - Bichat Hospital, Paris
  - Tenon Hospital, Paris

REFERENCES:
- [Result] Claessens YE, Debray MP, Tubach F, Brun AL, Rammaert B, Hausfater P, Naccache JM, Ray P, Choquet C, Carette MF, Mayaud C, Leport C, Duval X. Early Chest Computed Tomography Scan to Assist Diagnosis and Guide Treatment Decision for Suspected Community-acquired Pneumonia. Am J Respir Crit Care Med. 2015 Oct 15;192(8):974-82. doi: 10.1164/rccm.201501-0017OC. PMID 26168322
- [Result] Le Bel J, Hausfater P, Chenevier-Gobeaux C, Blanc FX, Benjoar M, Ficko C, Ray P, Choquet C, Duval X, Claessens YE; ESCAPED study group. Diagnostic accuracy of C-reactive protein and procalcitonin in suspected community-acquired pneumonia adults visiting emergency department and having a systematic thoracic CT scan. Crit Care. 2015 Oct 16;19:366. doi: 10.1186/s13054-015-1083-6. PMID 26472401
- [Result] Das D, Le Floch H, Houhou N, Epelboin L, Hausfater P, Khalil A, Ray P, Duval X, Claessens YE, Leport C; ESCAPED Study Group. Viruses detected by systematic multiplex polymerase chain reaction in adults with suspected community-acquired pneumonia attending emergency departments in France. Clin Microbiol Infect. 2015 Jun;21(6):608.e1-8. doi: 10.1016/j.cmi.2015.02.014. Epub 2015 Feb 20. PMID 25704448
- [Derived] Hofmeister J, Garin N, Montet X, Scheffler M, Platon A, Poletti PA, Stirnemann J, Debray MP, Claessens YE, Duval X, Prendki V. Validating the accuracy of deep learning for the diagnosis of pneumonia on chest x-ray against a robust multimodal reference diagnosis: a post hoc analysis of two prospective studies. Eur Radiol Exp. 2024 Feb 2;8(1):20. doi: 10.1186/s41747-023-00416-y. PMID 38302850
- [Derived] Tubiana S, Epelboin L, Casalino E, Naccache JM, Feydy A, Khalil A, Hausfater P, Duval X, Claessens YE; ESCAPED study group. Effect of diagnosis level of certainty on adherence to antibiotics' guidelines in ED patients with pneumonia: a post-hoc analysis of an interventional trial. Eur J Emerg Med. 2023 Apr 1;30(2):102-109. doi: 10.1097/MEJ.0000000000000954. Epub 2022 Jun 27. PMID 35758267
- [Derived] Le Bel J, Pelaccia T, Ray P, Mayaud C, Brun AL, Hausfater P, Casalino E, Benjoar M, Claessens YE, Duval X; ESCAPED study group. Impact of emergency physician experience on decision-making in patients with suspected community-acquired pneumonia and undergoing systematic thoracic CT scan. Emerg Med J. 2019 Aug;36(8):485-492. doi: 10.1136/emermed-2018-207842. Epub 2019 Jun 24. PMID 31239315